CLINICAL TRIAL: NCT01211106
Title: Integrated vs Sequential Treatment for PTSD and Addiction Among OEF/OIF Veterans
Brief Title: Integrated vs Sequential Treatment for PTSD and Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZDA1-03-W10
Record Dates: First submitted 2010-09-27; First posted 2010-09-29 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: PTSD; Substance Addiction
Keywords: Treatment; PTSD; Addiction
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Behavior, Addictive | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Integrated Conditions (Experimental): Motivational enhancement therapy for addiction is combined with Prolonged exposure therapy for PTSD from the beginning of treatment. Both are delivered by the same provider throughout treatment.
  Interventions: Behavioral: Prolonged Exposure; Behavioral: Motivational Enhancement Therapy
- Arm 2 Sequential therapy (Experimental): Motivational enhancement therapy for addiction is delivered in the first 4 weeks and only after the addiction is addressed is the Prolonged exposure therapy for PTSD started.
  Interventions: Behavioral: Prolonged Exposure; Behavioral: Motivational Enhancement Therapy

INTERVENTIONS:
Behavioral: Prolonged Exposure — Although almost every form of psychotherapy has been advocated for PTSD, all evidence-based psychotherapies for PTSD are CBT programs that include variants of exposure therapy (Prolonged Exposure), cognitive therapy (CT), stress inoculation training (SIT), eye movement desensitization and reprocessing (EMDR), or combinations of these procedures. Exposure therapy involves helping PTSD sufferers to gradually confront distressing trauma-related memories and reminders to facilitate successful emotional processing of the trauma memory and reduction of associated distress. Most exposure therapy programs include both imaginable confrontation with the traumatic memories and in vivo exposure to trauma reminders.
Behavioral: Motivational Enhancement Therapy — Motivational Interviewing (MI) is defined as a client-centered, directive method for enhancing intrinsic motivation to change by exploring and resolving ambivalence. MI is characterized by its spirit, which is defined as collaboration with the client, evocation of the client's own perceptions, goals, and values, and respect for the client's autonomy.

SUMMARY:
The investigators are examining different treatment strategies of helping patients with PTSD and addiction.

DETAILED DESCRIPTION:
The investigators hypothesize that Veterans in the integrated conditions will show greater reductions in substance abuse and PTSD symptom severity at the end of treatment and at 6 and 9 month follow-ups. The investigators further hypothesize that offering Veterans Prolonged Exposure (PE) at the onset of treatment in the integrated condition will leader to greater retention and satisfaction than in the sequential treatment design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Persian Gulf Era veterans between 18-65 years old. Older individuals are unlikely to have served in Iraq or Afghanistan.
* Current diagnosis of PTSD (symptom duration > 3 months) with clinically significant trauma-related symptoms, as indicated by a score of at least 50 on the PCL
* Current abuse or dependence on alcohol, stimulants such as cocaine, opioids, including prescription opioids or benzodiazepines. Subjects must report using on average at least 10 out of 30 days prior to signing consent. Of note: subjects can be abusing or dependent upon nicotine or marijuana but these will not be considered sufficient for inclusion
* Provides informed consent
* Speaks and reads English

Exclusion Criteria:

* Current suicidal or homicidal ideation with intent and/or plan that, in the judgment of the investigator, should be the focus of treatment
* Meets current DSM-IV criteria for bipolar affective disorder, schizophrenia or any psychotic disorder
* Has unstable or serious medical illness, including history of stroke, seizure disorder, or unstable cardiac disease
* History of moderate or severe traumatic brain injury (TBI)
* Participation in Prolonged Exposure Therapy in the last 6 months.
* Initiation of a new psychotherapy program in the last 2 months.
* Active participation in a formal addiction treatment program. Actively engaged is defined as any visit in the program in the prior month and pending future appointments for the treatment of addictions
* Change in psychotropic medication in the 1 month prior to treatment except for the use of oxazepam for alcohol detoxification or a taper of a previously used benzodiazepine.
* Therapeutic use of a benzodiazepine greater than the equivalent of more than 40 mg of diazepam (see chart) at the time of randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-02; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David W. Oslin, MD, Principal Investigator — Philadelphia VA Medical Center, Philadelphia, PA
Locations (2):
- United States (2):
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - Philadelphia VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alpert E, Kaplan A, Nelson D, Oslin DW, Polusny MA, Ingram EP, Kehle-Forbes SM. Clusters Based on Within-Treatment Symptom Trajectories as Predictors of Dropout in Treatment for Posttraumatic Stress Disorder and Substance Use Disorder. J Dual Diagn. 2024 Jun 6:1-21. doi: 10.1080/15504263.2024.2355953. Online ahead of print. PMID 38843038
- [Derived] Scott JC, Lynch KG, Cenkner DP, Kehle-Forbes SM, Polusny MA, Gur RC, Chen S, Foa EB, Oslin DW. Neurocognitive predictors of treatment outcomes in psychotherapy for comorbid PTSD and substance use disorders. J Consult Clin Psychol. 2021 Nov;89(11):937-946. doi: 10.1037/ccp0000693. PMID 34881912
- [Derived] Kehle-Forbes SM, Drapkin ML, Foa EB, Koffel E, Lynch KG, Polusny MA, Van Horn DH, Yusko DA, Charlesworth M, Blasco M, Oslin DW. Study design, interventions, and baseline characteristics for the Substance use and TRauma Intervention for VEterans (STRIVE) trial. Contemp Clin Trials. 2016 Sep;50:45-53. doi: 10.1016/j.cct.2016.07.017. Epub 2016 Jul 19. PMID 27444425

RESULTS

PARTICIPANT FLOW:
Groups:
- Integrated Care: Prolonged exposure treatment is combined with Motivational Enhancement therapy from the beginning of treatment.
- Sequential Treatment: Motivational enhancement therapy is started for the first 4 weeks and only after addressing addiction is prolonged exposure therapy begun.
Period: Overall Study
Arm/Group | Integrated Care | Sequential Treatment
Started | 95 | 88
Completed | 82 | 77
Not Completed | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Care | Sequential Treatment | Total
Number analyzed (Participants) | 95 | 88 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (13.1) | 43.8 (13.0) | 44.1 (13.0)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 90 | 79 | 169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 49 | 42 | 91
  White | 37 | 38 | 75
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 95 | 88 | 183
PTSD Checklist score [Mean (Standard Deviation); unit: units on a scale] — PTSD Checklist score is a standardized self-report rating scale for PTSD comprising 17 items that correspond to the key symptoms of PTSD. Respondents indicate how much they have been bothered by a symptom over the past month using a 5-point (1-5) scale, circling their responses. Responses range from 1 Not at All - 5 Extremely thus the total score ranges from 17 - 85. Lower scores are associated with less severity/symptoms.
  units on a scale | 62.5 (11.3) | 63.6 (10.3) | 63.0 (10.9)
Percent days of heavy drinking [Mean (Standard Deviation); unit: percent days heavy drinking] | 51.7 (29.5) | 56.0 (29.6) | 53.8 (29.6)

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptoms
Description: PTSD checklist (PCL), the PCL version used with the civilian PCL. The PCL is a standardized self-report rating scale for PTSD comprising 17 items that correspond to the key symptoms of PTSD. Respondents indicate how much they have been bothered by a symptom over the past month using a 5-point (1-5) scale, circling their responses. Responses range from 1 Not at All - 5 Extremely thus the total score ranges from 17 - 85. Lower scores are associated with less severity/symptoms.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1: Integrated Conditions: Motivational enhancement therapy combined with Prolonged Exposure therapy.
- Arm 2 Sequential Therapy: MET followed by Prolonged Exposure
Arm/Group | Arm 1: Integrated Conditions | Arm 2 Sequential Therapy
Number analyzed (Participants) | 82 | 77
units on a scale | 55.5 (17.6) | 54.1 (17.9)

2. Primary Outcome: Drinking Outcome
Description: Percent days of heavy drinking during the sixteen weeks. The percentage of days in which heavy drinking occurred ranges from 0 - 100% with lower days associated with better outcomes.
Time Frame: 16 weeks
Population: The number of subjects available for this measure are greater than the PTSD outcome as drinking outcomes can be obtained at anytime and thus some participants provided data at the post study evaluation.
Measure: Mean (Standard Deviation); unit: percent days ofheavy drinking
Arm/Group | Integrated Care | Sequential Treatment
Number analyzed (Participants) | 83 | 79
percent days ofheavy drinking | 48.8 (38.4) | 40.6 (34.6)

ADVERSE EVENTS:
Arm/Group | Integrated Care | Sequential Treatment
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/88
Other Adverse Events (participants affected / at risk) | 0/95 | 0/88

LIMITATIONS AND CAVEATS:
Both arms of the study were active treatments. There was no control conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No